CLINICAL TRIAL: NCT04498858
Title: To Promote Tobacco Free Life in the Dental Practice in France: Feasibility Study
Brief Title: To Promote Tobacco Free Life in the Dental Practice in France
Acronym: TOBAFREE-DP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/70
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Tobacco Cessation; Dental Practice
Keywords: Tobacco cessation; dental practice; dentists; nicotine replacement therapy; counselling
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient
  Interventions: Other: Patient interview

INTERVENTIONS:
Other: Patient interview — Patient will be interviewed :
  * tobacco consumption
  * reported question asked by the dentist about his/her tobacco consumption
  * presence and nature of reported advices given by the dentist
  * presence and nature of actions proposed by dentists for patients reporting tobacco consumption, including prescription of NRT
  * presence and nature of the actions carried out or envisaged by these patients, including - smoking cessation
  * contact with the general practioner
  * Fagerstrom score (2 questions)
  * demographic variables, age, sex, level of education
  * satisfaction

SUMMARY:
In France, 34% of the adult population is smoking every day. The links between smoking and the development of several chronic disorders is well established and smoking is directly implicated in most of the oral diseases such as cancers of the oral cavity. Thus, dentists have access to an area of the body that is actively affected and this gives them a central role in dispensing advice and support regarding smoking cessation.

Dentists often cite issues such as lack of time or education as a reason for why they do not offer support for smoking cessation. A brief intervention can increase smoking cessation by 30 to 100% (ie 1-3% in absolute value). The "5A" approach integrates and extends the brief intervention. It consists in Asking about smoking status, Advising smokers of the benefit of stopping, Assessing motivation to quit, Assisting smokers in their quit attempt, Arranging follow-up with stop-smoking services. For practitioners who do not have enough time, a "3A" approach might be acceptable (Ask, Advice and Act) by providing details of local stop smoking services and/or prescribing nicotine replacement therapy (NRT). This very brief advice can be delivered in less than one minute.

To investigators knowledge, the role of dentists in the French national tobacco-free program is not yet documented in France while since 2016, dentists can prescribe NRT with some products taken in charge by the French health insurance.

An intervention taking part in the continuing professional development will be developed so the dentists fell legitimate, motivated and competent to talk with their patients about their tobacco consumption and to assist them in their smoking cessation process. This intervention based on the 5/3A approach and prescription of NRT will include a specific training and provision of management kit, with communication tools and network for appropriate references.

Investigators hypothesize that 5/3A approach is feasible with adequate intervention in dental practices in France (dentists apply the approach to 90% of their patients) and that the format, the conditions, the barriers and the lever actions of its implementation are known.

DETAILED DESCRIPTION:
In Europe, 29% of individuals are smokers, and tobacco use is directly related to 650,000 mortalities each year across the continent, around 14% of all deaths. In France, 34% of the adult population is smoking everyday (www.OFDT.fr). The links between smoking and the development of several chronic disorders is well established and long-term smokers are more likely to die from a disease directly related to their habit. Smoking is also responsible for a large burden of evitable morbidity.

From a dental perspective, smoking is directly implicated in most of the oral diseases (periodontal diseases, dermatological disorders of the oral mucosa, bad breath, peri-implantitis…). Smoking is also directly related to the development of potential malignant lesions of the oral mucosa and cancer of the oral cavity. Thus, dentists have access to an area of the body that is actively affected and this gives them a central role in dispensing advice and support regarding smoking cessation. Fifty percent of the EU population regularly visit a dentist and in France, a survey conducted in 2014 showed that 63.5 % of the 15-75 year-old respondents reported to have visited their dentist in the 12 previous months. These data show that dentists have access to a large number of smokers with the opportunity to offer information and support regarding smoking cessation.

Dentists often cite several issues, such as lack of time or limited education, to explain why they do not offer support for smoking cessation. A Cochrane review showed that a brief intervention by health professionals is effective in helping tobacco users to quit. This 'brief' advice in primary care settings has been shown to increase smoking cessation by 1-3%. Whilst this number seems small, it represents a large number of people from a population point of view. By referring to stop smoking services, successful cessation increased to 15%.

The "5A" approach to smoking cessation is the internationally accepted approach integrating a "brief intervention" for nicotine users. The 5A protocol can be summarized as follows:

* Ask about and record smoking status.
* Advise smokers of the benefit of stopping in a personalized and appropriate way.
* Assess motivation to quit (using stages of change model).
* Assist smokers in their quit attempt.
* Arrange follow-up with stop smoking services.

Advice from the healthcare practitioner does not have to be focused on the details of cessation and requires only three minutes. Whilst knowledge of the treatment modalities to result in cessation are useful, ultimately the specialized stop-smoking services will be able to discuss any potential issues adequately with the individual.

For practitioners who genuinely do not have time, a 3A approach may be acceptable. As dentists seem to be content with the first two 'A' in either scenario, it is the addition of 'action' on responses which increases success rates in quitting. This can be summarized as follows:

* Ask and record smoking status.
* Advise patient of personal health benefits.
* Act on patient's response by providing details of local stop smoking services and/or prescribing NRT.

This very brief advice can be delivered in less than one minute and there is an absence of conclusive evidence to indicate that the 5A approach is more successful than the 3A.

The authors are aware of the need to be pragmatic in the approach to smoking cessation in the dental setting, therefore advice that the 3A approach is the best brief intervention to be undertaken by dentists. It is easier to complete than the 5A and, if done properly, both approaches result in similar rates of smoking cessation. Dentists can choose the most convenient approach to their practice and refer their patients to specialized care when needed.

In a recent study, the effectiveness of a very brief structured counselling for tobacco was evaluated cessation in Swedish dental clinics. It was observed that a brief and structured counselling based on the 5A model in dental practice may achieve positive behavioural modifications among tobacco users, with significant reduction of tobacco consumption.

General dentists are used to deliver preventive messages focused on oral hygiene (tooth brushing, flossing, reduction of sugar intake…) but they are less likely to deliver general health-promoting messages. A literature review on the factors associated with the delivery of lifestyle support in general dental practice has shown that organizational changes in dental practices to encourage more team working and professional time for lifestyle support may influence delivery of such messages. It was also observed that dental professionals who are smokers may require training to develop their beliefs about the effectiveness of smoking cessation interventions.

Thus, even if they are well positioned to offer tobacco cessation advice and support, dentists do not always discuss their patient's tobacco use. A study by Smith et al showed that motivated dentists were particularly good at offering smoking cessation to patients. However, less than 50% of dental practices involved in the study offered referrals to stop smoking services. Further studies confirm that dentists are often poor at referring to stop smoking services, or offering brief interventions at the dental practice. There is therefore a need to understand the factors, barriers and lever action which influence dentists 'practices toward tobacco cessation advice and support. When it is considered that patients expect their oral health professionals to assist in cessation attempts, this gives further reason for dental professionals to understand and implement cessation techniques.

By utilizing the 'stages of change' approach to smoking cessation, an individual's willingness to quit smoking can be ascertained, with provision of knowledge on potential interventions empowering patients to make their own decisions on cessation modalities. Since 2016, in France, dentists can prescribe nicotine replacement therapy (NRT) and it will be reimbursed to the patients by the French health insurance at a rate of 65%. NRT can reduce physical cravings and pharmacotherapies can reduce the desire to smoke. Stop-smoking services can provide smokers with interpersonal support and electronic cigarettes are increasing in popularity but cannot be recommended as a completely safe way of delivering nicotine. Interpersonal support in combination with NRT and/or pharmacotherapy is now considered the safest and most successful method of smoking cessation.

To our knowledge, the role of dentists in the French national tobacco free program is not yet documented in France while the "Conseil de l'Ordre des Chirurgiens-dentistes" was associated to this program launched in 2014. Also, the role of dentists was underlined in the HAS recommendations in 2014 as any other health professional.

Because of the impact of tobacco smoking on oral health and the frequency of individuals visiting them, dentists should be made aware and feel legitimate in their first line role in terms of smokers 'management combining 5/3 A approach, prescription of NRT and reference to specialized care.

Continuous professional training is mandatory and could be an opportunity to improve dentists 'motivation and skills to provide advice and support to their patients. By familiarizing the dental team with gold-standard cessation interpersonal and NRT support and by providing them with appropriate communication and reference resources, it can be ensured that smokers are assisted at every available opportunity.

The idea is to develop an intervention that take part in the quality approach of the dental practice in the context of the continuing professional development so the dentists fell motivated, legitimate and competent to talk with their patients about their tobacco consumption and to assist them in their smoking cessation process. This intervention based on the 5/3A approach and prescription of NRT will include adequate training and provision of management kit with communication tools and network for appropriate references. To develop this intervention, it is necessary to have a comprehensive acknowledgement of all the factors with which the intervention fits, relative to the recommendations, to the health professional him/herself, the human and organizational environment.

Investigators hypothesize that 5/3A approach is feasible in dental practices in France (dentists apply the approach to 90% of their patients) with adequate intervention and that the format, the conditions, the barriers and the lever actions of its implementation are known.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* smoker
* Will to participate to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of trained dentists to 3/5A strategy
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
5/3A approach | 1 month after inclusion (day0)
  Acceptability for performing the 5/3A approach in the dental practice

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided